CLINICAL TRIAL: NCT03620214
Title: Descriptive Study of the Physiological and Oral Parameters of the Young Child to the Adolescent
Brief Title: Physiological and Oral Dental Parameters of Young Child
Acronym: PhyDentchild
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18043
Record Dates: First submitted 2018-03-28; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Odontology
Keywords: CHILD; GROWTH; PHYSIOLOGICAL PARAMETERS; FACE; MAXILLARY

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy children: Healthy children consulting at the odontology department of Reims CHU for carious screening or orthodontic diagnosis; excluding research

SUMMARY:
The aim of this study is to measure some oral and maxillofacial physiological parameters, with a view to creating a modular prototype articulator from young children to adolescents by 3D printing.

DETAILED DESCRIPTION:
In the dental field, the articulators present different interests during the diagnostic and treatments of the dental diseases. Thus they are used to perform dental prostheses, pre-orthodontic analysis or in the context of dysfunction of the manducatory apparatus.

Many children affecting with genetic disease need prosthetic rehabilitation. However, none commercial articulators are adaptable to children. Consequently little dental prosthetic are taken before adolescence, or even adulthood.

The aim of this study is to measure some oral and maxillofacial physiological parameters, with a view to creating a modular prototype articulator from young children to adolescents by 3D printing.

On average, 30 children per week visit the dental department of Reims CHU for dental screening or orthodontic diagnosis. From this cohort, an epidemiological study will be carried out. It will concern different physiological parameters of the face and the oral cavity necessary to make a prototype articulator.

Ideally, the creation of a modular articulator to monitor the growth of a child would remove a number of diagnostic locks, therapeutic and technical.

ELIGIBILITY:
Inclusion Criteria:

First 30 children in each age group ([3; 6 [; [6; 9 [; [9; 12]) presenting to the Odontology Division as part of a first dental care or orthodontic consultation.

Exclusion Criteria:

* Any child consulting to the Odontology Department in emergencies.
* Any child coming out of the weight-of- height growth curve. For example, a child below is considered to have hypo-development. Conversely, a child located above the growth curve is considered to be hyper-developed.
* Any child with absence of at least 2 teeth per quadrant whether it is a genetic etiology (agenesis), infectious (avulsion) or traumatic (expulsion).
* Any child with a maxillofacial malformation generating disorders of the face development (ex: child with a cleft palate ...)
* Any child presenting a Class III of Angle. Indeed the intermaxillary ratios being reversed, a hypo-development of the maxillary is often observed.
* Any child with a cognitive impairment that limits the understanding of the examination undertaken.
* Any non-cooperating child

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy children consulting at the odontology department of Reims CHU for carious screening or orthodontic diagnosis; excluding research
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-09-23 (Estimated); Study Completion 2018-09-23 (Estimated)

PRIMARY OUTCOMES:
Inter-ear distance | Day 0
  distance between ears
Measurements of the upper floor of the face | Day 0
  distance between the hair line and the glabella (in cm) measured using a calliper
Inter-commissural distance when closed and opened mouth | Day 0
  Distance between commissures of the lips, mouth opened and closed
Tempo-mandibular joint | Day 0
  The calculation of the condylar track inclination (in degrees) will be done using an axiographe or the displacement of the mandible in propulsion
Frontal plane | Day 0
  distance between the two pterygoid-maxillary ligaments
Inter canine distance | Day 0
  distance between canines
Measurements of the middle floor of the face | Day 0
  distance between the glabella and the sub nasal point (in cm) measured using a calliper
Measurements of the lower floor of the face | Day 0
  distance between the sub nasal point ans the chin (in cm) measured using a calliper

SECONDARY OUTCOMES:
age | Day 0
  age in years
sex | Day 0
  male or female

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France